CLINICAL TRIAL: NCT00222287
Title: The Effect of Feldenkrais Lessons on Walking and Balance
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Melbourne (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC No. 040730; NCT00222313 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-22 (Estimated); Status verified 2006-09

CONDITIONS: Accidental Falls; Exercise
Keywords: Feldenkrais Method; movement class; balance; Four square step test; Activities Specific Balance Confidence Scale; systems theory
MeSH Terms: conditions — Motor Activity

INTERVENTIONS:
Behavioral: Feldenkrais Movement class

SUMMARY:
The purpose of this study is to investigate the effects of a series of Feldenkrais movement lessons on mobility and balance, particularly for older adults. The investigators hypothesise that mobility and balance will improve following the classes.

DETAILED DESCRIPTION:
The Feldenkrais Method is an educational process which involves exploration of novel movement sequences that lead to expansion of the movement repertoire. This Method has been used with the aim of improving balance and mobility in several studies, and has been compared to the benefits of Tai Chi for improving balance in older adults. The current study investigates the effects of a 10 week series of Feldenkrais movement classes on gait parameters as measured on an instrumented gait mat, a balance test of stepping and turning (the Four Square Step Test) and a questionnaire about balance confidence (the Activites Specific Balance Confidence scale.

ELIGIBILITY:
Inclusion Criteria:

* community dwelling older adults (aged over 65)
* able to independently ambulate indoors and outdoors

Exclusion Criteria:

* currently undergoing physiotherapy treatment
* unable to comprehend written english
* unable to give informed consent
* walking with a walking frame indoors

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2005-12

PRIMARY OUTCOMES:
Balance Confidence (as measured by ABC scale)
Tempo-spatial parameters of gait
Time to complete Four Square Step Test

CONTACTS AND LOCATIONS:
Overall Officials: Mary Galea, PhD, B App Sc (PT), Study Director — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia